CLINICAL TRIAL: NCT06180941
Title: The Effect of Magnesium Sulfate in Comparison to Clonidine as Adjuvants to Bupivacaine 0.25% in Supraclavicular Brachial Plexus Block in Pediatric Upper Limb Surgeries. Prospective, Randomized, Double-blind Study
Brief Title: Adjuvants for Bupivacaine in Brachial Plexus Block in Pediatrics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Abdulbassit mohammed abdou, residant physician, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: brachial plexus block.
Record Dates: First submitted 2023-11-21; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Upper Limb Injury
MeSH Terms: conditions — Arm Injuries | interventions — Magnesium Sulfate; Clonidine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnesium sulfate as adjuvant to bupivacaine. (Active Comparator): Group M: 2mg/kg Magnesium sulfate will be added to 0.5 mL.kg-1 of 0.25% bupivacaine (max 2 mg/kg) with a total volume of 0.5 ml/kg, (according to the spread of local anesthetic surrounding the brachial plexus)
  Interventions: Drug: magnesium sulfate.
- clonidine as adjuvant to bupivacaine. (Active Comparator): Group C: 0.75 μg.kg-1 of clonidine will be added to 0.5 mL.kg-1 of 0.25% bupivacaine (max 2 mg/kg) with a total volume of 0.5 ml/kg, (according to the spread of local anesthetic surrounding the brachial plexus)
  Interventions: Drug: clonidine.

INTERVENTIONS:
Drug: magnesium sulfate. — magnesium sulfate as adjuvant to bupivacaine in supraclavicular brachial plexus block in pediatrics.
  Arms: magnesium sulfate as adjuvant to bupivacaine.
Drug: clonidine. — clonidine as adjuvant to bupivacaine in supraclavicular brachial plexus block in pediatrics.
  Arms: clonidine as adjuvant to bupivacaine.

SUMMARY:
Among paediatrics aging 3:12 who are going to have upper limb surgery,does adding clonidine to bupivacaine improve brachial plexus block outcome in comparison with magnesium sulfate with bupivacaine?

DETAILED DESCRIPTION:
In upper extremity surgery, brachial plexus blocks are often preferred due to their advantages, such as long postoperative analgesic efficacy and shortening the length of hospital stay. This application reduces the use of opioids for postoperative analgesia and provides protection from their side effects. However, procedure failure, nerve injury and intravascular injection are the most common complications in the past years. In recent years, performing ultrasound-guided blocks has increased the success of the procedure and decreased the complication rate. Low number of studies, knowledge and experience in paediatric patients led to worries that complications will be more common and caused less use of regional techniques. However, good visualization of the anatomy in ultrasound-guided blocks and successful results in adult patients brought up the application of ultrasound-guided brachial plexus blocks in children.

Effective postoperative analgesia improves patient's outcome in terms of early ambulation, decreased complications, and reduced incidence of postoperative chronic pain. Regional anaesthetics is a safe and effective method for upper limb surgeries. This method can prolong analgesia and reduce postoperative pain. Nowadays, peripheral nerve block has found an important role in anaesthesiology. Safety and high success rate have made it a common technique in outpatient and inpatient anaesthetics. Upper limb surgeries are mostly performed under peripheral nerve blocks such as brachial plexus block. Brachial plexus may be blocked in the level above the clavicle as interscalene and supraclavicular blocks or below the clavicle as infraclavicular and axillary blocks. Supraclavicular brachial plexus block is used for surgeries of the upper limb below the arm, from elbow to hand. Brachial plexus is blocked in the level between trunks and divisions. In this level, a small volume of local anaesthetic is needed for reliable block. The guide of ultrasound allows the anaesthesiologist to see the subclavian artery as a bold marker and neural structures around it above the 1st rib Regional anaesthetics may be one of the best solutions for intraoperative and postoperative paediatric pain management; Supraclavicular brachial plexus block is considered as one of the most effective anaesthetic methods for upper extremity surgeries. Its major drawback, especially in children, is the risk of pneumothorax, vascular puncture, and failure of the procedure due to inaccurate placement of the needle. Ultrasound-guided needle placement may reduce the risk of complications and increase the accuracy of block, particularly in paediatric patients. According to the surgeon's preference and due to the need for a tourniquet at the proximal part of the humerus in all surgeries regardless of the type of surgery, we considered supraclavicular block to be more suitable than more distal ones. This block can be done with only one injection around the plexus and provides sufficient anaesthetics at the tourniquet site as well.

Lignocaine and bupivacaine are the commonly used local anaesthetics in Brachial plexus blocks. Lidocaine is an aminoamide, moderate acting local anaesthetic that blocks the peripheral afferents acting on voltage-dependent sodium channels, Bupivacaine is a potent local anaesthetic with unique characteristics from the amide group of local anaesthetics, which was first discovered in 1957 and widely used for prolonged local and regional anaesthetics.

To increase the duration of local anaesthetic effect in the supraclavicular block,Local anaesthetics provide good anaesthetics in regional blocks, but have shorter duration of postoperative analgesia. Thereby, various adjuncts like opioids, clonidine, neostigmine, dexamethasone, alpha-2 agonists, dexmedetomidine, ketorolac, ketamine, and low-level laser therapy, have been used in regional blocks to achieve desirable analgesia.

In the meantime, epinephrine is mostly used. Although epinephrine reduces the absorption of local anaesthetics, reduces their toxicity, and prolongs anaesthetic duration, it can cause hypertension and tachycardia. Therefore, its usage is limited when the patients have cardiovascular disease or hyperthyroidism Magnesium sulphate is an N-methyl D-aspartate (NMDA) receptor antagonist in the central nervous system (CNS) and peripheral nervous system (PNS). The NMDA receptor complex contains binding sites for antagonists such as magnesium. Magnesium is used as an adjuvant in peripheral nerve block. Anti-nociceptive effects of magnesium are due to the regulation of calcium influx into the cell and antagonism of the NMDA receptors. Many clinical studies have demonstrated that magnesium used during general anaesthetics reduced anaesthetic requirement and postoperative rescue analgesic. Magnesium has been commonly used as an antihypertensive agent. Magnesium may prevent postoperative shivering. More recently, it has been shown that magnesium sulfate decreased the effects of aminoamide local anaesthetics on rat sciatic nerves in vivo.

Recently, alpha-2 receptor-stimulating drugs due to excellent sedative effects, analgesia, and anaesthetics with hemodynamic stability have been considered These pharmacologic properties have been employed clinically to achieve the desired effects in regional anaesthetics.

Clonidine, an a2 adrenergic agonist has sedative, analgesic, perioperative sympatholytic with cardiovascular stabilizing effects and has been tried in combination with local anaesthetic drugs to enhance regional anaesthetics.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists Classes I and II patients.
* within the age group of 3-12 years.
* requiring unilateral upper limb surgery at or below the elbow.

Exclusion Criteria:

* The patients that have contraindications to regional anaesthetics, previous nerve injuries, history of allergy to study drugs, history of bleeding disorders.
* children with any mental disability which will confound pain assessment or inability to understand the pain scale used in the study.
* patients on anticoagulants.
* patients with any major systemic illness will be excluded from the study.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Time to first rescue analgesia. | 24 hours
  The time(in hours) to first rescue analgesia which is defined as the time since the block performance till the first administration of any rescue analgesia in the postoperative period.

SECONDARY OUTCOMES:
Postoperative analgesia. | 24 hours
  Wong-Baker faces pain rating scale (WBFPS) will be used for pain assessment in both the groups at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 12 h, and 24 h. The number of children with WBFPS >6 at any time point will be recorded for both groups.
  Wong-Baker faces pain rating scale (WBFPS) presents 6 faces with increasing degree of pain from left to right. Each face is attributed scale from 0 to 10 indicated on scale. Children will be asked to choose the face that best describes his or her own pain.